CLINICAL TRIAL: NCT00438776
Title: Safety and Efficacy Trial of Olanzapine in Outpatients With Pathological Gambling
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Eli Lilly and Company (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F1D-US-X165
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Pathological Gambling
MeSH Terms: conditions — Gambling | interventions — Olanzapine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- olanzapine (Active Comparator): active zyprexa (olanzapine)
  Interventions: Drug: olanzapine
- sugar pill (Placebo Comparator): Placebo (fake pill)
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: olanzapine — 2.5mg to 15mg daily
  Other Names: zyprexa
  Arms: olanzapine
Drug: sugar pill — matching placebo to olanzapine
  Other Names: fake pill
  Arms: sugar pill

SUMMARY:
The purpose of this research study is to evaluate the efficacy (effectiveness) and safety of olanzapine in treating pathological gambling.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients aged 18- 75 years of age.
2. Patients will have problematic gambling behavior of at least 6 months duration that meets the DSM-IV definition of pathological gambling and a South Oaks Gambling Screen Score greater than 5.
3. All patients will have a complete medical and psychiatric history, physical examination, laboratories, and ECG before study entry.
4. Baseline laboratory values and ECG must be normal, or abnormalities must be clinically insignificant.
5. Patients will not have received any psychotropic medication for at least one week prior to the first study visit.

Exclusion Criteria:

1. Patients who have any significant and/or unstable gastrointestinal, neurological, endocrine, cardiovascular, pulmonary, renal, hepatic, immunological or hematological disease; organic brain disease; or cancer as determined by history, physical, ECG, and laboratory examination.
2. Patients who are pregnant, intending to become pregnant, nursing, at risk for pregnancy, or not practicing medically acceptable birth control. (A blood pregnancy test will be performed at the screening visit).
3. Patients who have ever had psychotic symptoms, who have ever met DSM-IV criteria for a manic episode (i.e., have bipolar I disorder), or who have met criteria for DSM-IV psychoactive substance dependence in the past 1 month.
4. Patients who meet DSM-IV criteria for antisocial or borderline personality disorder.
5. Patients who use any medications which, in the judgment of the investigator, might have psychotropic effects, or interact unfavorably with olanzapine. For example, patients taking diet pills or stimulants will not be enrolled.
6. Patients who have taken any psychiatric medication within 7 days prior to the screening assessment.
7. Patients who have a history of hypersensitivity to olanzapine.
8. Patients who display clinically significant suicidal ideation.
9. Patients who have recently (within the past 3 months) begun any type of non-pharmacologic treatment for pathological gambling (including psychotherapy, behavior therapy, group therapy, or family therapy). This does not exclude participation in support groups (e.g., Gamblers Anonymous.) Patients who have been involved in long-standing psychological therapies (e.g., psychotherapy for at least the last 3 months) will be permitted to continue in that therapy provided that no new therapeutic technique or increase in frequency of psychotherapy occurs concurrent with the study.
10. Patients who exhibit or suggest that they may display behavior that will not be conducive to the study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pathological Gambling Adaptation of the Yale-Brown Obsessive Compulsive Scale (PG-YBOCS) | per protocol

CONTACTS AND LOCATIONS:
Overall Officials: Susan L McElroy, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] McElroy SL, Nelson EB, Welge JA, Kaehler L, Keck PE Jr. Olanzapine in the treatment of pathological gambling: a negative randomized placebo-controlled trial. J Clin Psychiatry. 2008 Mar;69(3):433-40. doi: 10.4088/jcp.v69n0314. PMID 18251624